CLINICAL TRIAL: NCT03641404
Title: Pilot Study to Investigate the Efficacy of Ergothioneine to Delay Cognitive Decline in Mild Cognitively Impaired Subjects
Brief Title: Investigating the Efficacy of Ergothioneine to Delay Cognitive Decline (Pilot)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Collaborators: National University of Singapore (Other); National University Health System, Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2017/00982; 1823117J (Clinical Trial No.) (Other: Health Science Authority (Singapore))
Record Dates: First submitted 2018-07-16; First posted 2018-08-22 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2018-05

CONDITIONS: Mild Cognitive Impairment
Keywords: ergothioneine; mild cognitive impairment; dementia; dietary antioxidant
MeSH Terms: conditions — Cognitive Dysfunction; Dementia | interventions — Ergothioneine

STUDY DESIGN:
Intervention Model Description: Randomized, double-blinded, placebo-controlled study
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Investigational compound and placebo coded by manufacturer. Codes provided in envelope will only be unsealed at the end of the study (data assessment) or in case of emergency.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ergothioneine (Active Comparator): Subjects will consume 25mg ergothioneine (capsule), 3 times weekly (Monday, Wednesday, and Friday) for a total of 52 weeks.
  Interventions: Drug: L-ergothioneine
- Placebo (Placebo Comparator): Subjects will be given placebo (99% microcrystalline cellulose, 1% magnesium stearate; capsule), 3 times weekly (Monday, Wednesday, and Friday) for a total of 52 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: L-ergothioneine — Ergothioneine is naturally occurring thiol compound obtained solely from diet in humans. Ergothioneine is widely reported to be a natural antioxidant and anti-inflammatory compound. In addition we hypothesize that this compound will be beneficial in improving cognition.
  Arms: Ergothioneine
Drug: Placebo — Placebo. Study control (99% microcrystalline cellulose, 1% magnesium stearate)
  Arms: Placebo

SUMMARY:
With the growing burden of dementia (including Alzheimer's disease), and the lack of efficacious therapies, there is an urgent need to identify new therapeutics.

Ergothioneine (ET) is a naturally occurring thiol derivative of histidine, obtained solely through diet and is able to accumulate in the body and brain, through the action of a specific transporter, OCTN1. In addition to a wide variety of in vitro and in vivo (animal) studies demonstrating the antioxidant, anti-inflammatory properties of ET, several studies have demonstrated the neuroprotective potential of ET in various cell and animal models.

Based on the ability of ET to counteract the underlying pathology of AD dementia, it is hypothesize that ET supplementation may prevent cognitive decline, especially in individuals at risk of cognitive impairment. This will be assessed using a randomized, double blinded, placebo-controlled, intervention study to test the ability of ET to delay or reverse cognitive impairment in elderly individuals with mild cognitive impairment.

DETAILED DESCRIPTION:
Ergothioneine (ET) is a naturally occurring thiol/thione obtained in humans solely through diet. It is able to accumulate in specific cells and tissues (including the brain), via a specific transporter, OCTN1, at high levels. Although the exact physiological function(s) of ET have yet to be elucidated, numerous reports have demonstrated that this compound can scavenge reactive oxygen species (such as hydroxyl radicals, hypochlorous acid, and peroxynitrite), modulate inflammation, and chelate divalent metal ions. These processes are all implicated in the pathology of dementia. Various studies in cell and animal models have also highlighted the potential neuroprotective capabilities of ET following insult by various neurotoxic agents such as cisplatin and amyloid beta peptide.

Studies demonstrated that ET dose-dependently protected PC12 cells against beta amyloid-induced apoptotic death, and later was shown to protect against neuronal injury caused by direct administration of amyloid beta into the mouse hippocampus, thereby increasing scores in active avoidance and water maze tests. ET also dose-dependently extend lifespan of a transgenic Caenorhabditis elegans model of AD by reducing amyloid oligomer formation. Other studies also demonstrated that ET is also able to attenuate oxidative stress and prevents cognitive deficits in a D-galactose-induced dementia mouse model; protect against N-methyl-D-aspartate-induced cytotoxicity in rat retinal neurons; and prevent cisplatin-induced neuronal damage in cell cultures and mice.

To date no studies have evaluated the therapeutic ability of ET, clinically, to delay or halt cognitive decline. Prior studies administering pure ET to humans provide insights into the pharmacokinetics and demonstrate the safety of this compound, laying the foundations for this clinical study. The present proposal will shed light onto a relatively lesser known natural compound and the therapeutic capabilities it possesses, which has the potential to significantly impact the economic and societal burdens of dementia.

ELIGIBILITY:
Inclusion Criteria:

* Elderly individuals 60 - 90 years of age
* Chinese ethnicity (from other local cohort studies)
* Demonstrate amnestic mild cognitive impairment (assessed by panel of psychiatrists)
* Independent and able to travel to study site without assistance
* No other severe underlying conditions or terminal illnesses
* Capable of understanding the study and requirements and able to provide informed consent to participate
* Willing to commit to the year-long study, comply with study administration and periodic blood and urine sampling

Exclusion Criteria:

* Inability to understand the risks and requirements of the study for any reason
* Any intolerance to lactose, and/or allergies to mushrooms
* History of cardiovascular complications, diabetes, hypertension or hypercholesterolemia, or other pre-existing condition that may prevent them from completing the study
* Evidence of anaemia or other significant haematological conditions
* History or mental illness, depression or other underlying psychiatric illnesses
* History of drug or alcohol abuse
* Involvement in another study requiring administration of an investigational compound in the past 30 days
* Subjects whose blood analysis reveal and extremes of liver or kidney function markers (from baseline screening)
* Deemed unfit for any reason as determined by the principal/co-investigator

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Demonstrating uptake of ergothioneine following dietary supplementation | 12 months
  This pilot study will evaluate the ability of oral ergothioneine supplementation to raise levels of ergothioneine in the body (blood measurements) over the one year period
Demonstrate safety of oral ergothioneine supplementation | 12 months
  This study will evaluate the safety oral ergothioneine supplementation over a period of 12 months. Safety is monitored through monthly visits (assessment and feedback on adverse reactions) and quarterly blood assessment (blood counts, liver and renal function).
Evaluating the impact of ergothioneine supplementation to modulate oxidative damage | Over 12 months
  The ability of oral ergothioneine supplementation to modulate oxidative stress in the subjects will be assessed through changes in plasma and urinary oxidative damage biomarkers collected at baseline and quarterly (every 3 months) over the 12-month study duration.
Evaluate the impact of ergothioneine supplementation to modulate inflammation | Over 12 months
  The ability of oral ergothioneine supplementation to modulate inflammatory status in the subjects will be assessed through measurement of inflammatory cytokines in the plasma at baseline and quarterly (every 3 months) over the 12-month study duration.

SECONDARY OUTCOMES:
Assessment of plasma neurofilament light chain (NfL) protein levels | 12 months (assessed at baseline and every 3 months)
  Elevated levels of NfL are suggested to be a biomarker of neurodegeneration and hence changes in this biomarker could reflect pathological changes. Increasing levels of NfL suggest progression or increasing severity of neurodegeneration and cognitive impairment whereas unchanged or decreasing levels of NfL may indicate a stabilisation or mitigation of neurodegeneration.
Evaluation of cognition using the Singapore Modified - Mini Mental State Examination Scores (Cognitive function assessment) | 12 months (assessed baseline, 6 months and 12 months)
  30 point questionnaire to assess for cognitive function and memory recall, with a minimum score of 0 and maximum of 30; where higher is better. A score of less than 7 may be indicative of cognitive impairment.
Evaluation of dementia stage using the Clinical Dementia Rating Scale (CDR). | 12 months (assessed baseline, 6 months and 12 months)
  CDR evaluates multiple domains including memory, orientation, judgement and problem solving, home and hobbies, community and personal care using a 5-point scale (0, 0.5, 1, 2, 3, where higher score indicates increasing severity of dementia) from 0 (no dementia) to a maximum of 3 (severe dementia). A 0.5-1 score indicates possible to mild cognitive impairment.
Neuropsychological test battery: Rey Auditory Verbal Learning Test (Cognitive function assessment) | 12 months (assessed baseline, 6 months and 12 months)
  The Rey Auditory Verbal Learning Test (RAVLT) evaluates short-term auditory-verbal memory, rate of learning, learning strategies, retroactive, and proactive interference, presence of confabulation of confusion in memory processes, retention of information, and differences between learning and retrieval. Participants are given a list of 15 unrelated words repeated over five different trials and are asked to repeat the words. Another list of 15 unrelated words are given and the client must again repeat the original list of 15 words and then again after 30 minutes. A score out of 75 for immediate recall and 30 for secondary and delayed recall, whereby higher indicates better verbal learning and memory.
Neuropsychological assessment battery: Digit Span test (Cognitive function assessments) | 12 months (assessed baseline, 6 months and 12 months)
  The digit span task is a measure of working memory, based on a person's ability to recall a sequence of numerical digits evaluating short-term and working memory. A maximum score of 16 for forward and 14 for backward where higher indicates score indicates better short-term and working memory and cognitive control.
Neuropsychological assessment battery: Block Design Test (Cognitive function assessment) | 12 months (assessed baseline, 6 months and 12 months)
  The block design test examines the spatial visualisation ability and motor skills of an individual where the subject is asked to replicate a different design patterns using cubes. Scoring as based on timing and correct pattern with a maximum score of 68 with higher indicating better spatial visualisation.
Neuropsychological assessment battery: Symbol Digit Modality Test scores (Cognitive function assessment) | 12 months (assessed baseline, 6 months and 12 months)
  The symbol digit modality is a cognitive assessment test for evaluating information processing speed and attention. Increased written and oral symbol score (1 point per correct answer, minimum of 0 and maximum of 100 limited by the test form) over 90 seconds indicates better processing speed.
Neuropsychological assessment battery: Semantic Verbal Fluency Test (Cognitive function assessment) | 12 months (assessed baseline, 6 months and 12 months)
  The Semantic Verbal Task involves asking the subject to name as many animals (part 1) and fruits (part 2) as they can in 60 seconds, which each correct answer adding one point. Scores are tallied from parts 1 and 2, with higher scores (no limit, only based on time) indicating better language, semantic memory, and processing ability.
Neuropsychological assessment battery: Colour Trials Test (Cognitive function assessments) | 12 months (assessed baseline, 6 months and 12 months)
  The colour trails test assesses sustained and dividend attention, and executive function involving parts 1 - connecting numbered circles in sequence and part 2 - requires alternating between circles of different colours (pink and yellow) while connecting them in numerical order. The time taken to complete parts 1 and 2 are recorded (as well as errors) with faster time indicating better attention and cognitive flexibility.
Evaluation of Geriatric Anxiety Inventory (Neuropsycological assessment) | 12 months (assessed baseline, 6 months and 12 months)
  The geriatric anxiety inventory is a self-reported assessment to identify anxiety syndromes in elderly individuals, through a series of 20 questions (with minimum of 0 and maximum score of 20) with a higher score indicating the possibility of underlying anxiety and greater than 9 indicating the possibility of an underlying anxiety disorder. At the conclusion of the study a reduction or absence of change is expected in the geriatric anxiety score.
Evaluation of Geriatric Depression Scale (Neuropsycological assessment) | 12 months (assessed baseline, 6 months and 12 months)
  The geriatric depression scale is a self-reported assessment to identify depressive symptoms in elderly individuals, through a series of 15 guided questions (with minimum of 0 and maximum score of 15) with a higher score indicating greater severity and greater than 5 indicating the possibility of an underlying depressive syndromes. At the conclusion of the study a reduction or absence of change is expected in the geriatric depression scale.

CONTACTS AND LOCATIONS:
Overall Officials: Rathi Mahendran, Principal Investigator — National University of Singapore; Barry Halliwell, Principal Investigator — National University of Singapore; Christopher Chen, Principal Investigator — National University Hospital, Singapore
Locations (1):
- National University Cancer Institute, Singapore, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Halliwell B, Cheah IK, Tang RMY. Ergothioneine - a diet-derived antioxidant with therapeutic potential. FEBS Lett. 2018 Oct;592(20):3357-3366. doi: 10.1002/1873-3468.13123. Epub 2018 Jun 15. PMID 29851075
- [Background] Cheah IK, Halliwell B. Ergothioneine; antioxidant potential, physiological function and role in disease. Biochim Biophys Acta. 2012 May;1822(5):784-93. doi: 10.1016/j.bbadis.2011.09.017. Epub 2011 Oct 4. PMID 22001064
- [Background] Halliwell B, Cheah IK, Drum CL. Ergothioneine, an adaptive antioxidant for the protection of injured tissues? A hypothesis. Biochem Biophys Res Commun. 2016 Feb 5;470(2):245-250. doi: 10.1016/j.bbrc.2015.12.124. Epub 2016 Jan 6. PMID 26772879
- [Background] Cheah IK, Feng L, Tang RMY, Lim KHC, Halliwell B. Ergothioneine levels in an elderly population decrease with age and incidence of cognitive decline; a risk factor for neurodegeneration? Biochem Biophys Res Commun. 2016 Sep 9;478(1):162-167. doi: 10.1016/j.bbrc.2016.07.074. Epub 2016 Jul 19. PMID 27444382
- [Background] Cheah IK, Tang RM, Yew TS, Lim KH, Halliwell B. Administration of Pure Ergothioneine to Healthy Human Subjects: Uptake, Metabolism, and Effects on Biomarkers of Oxidative Damage and Inflammation. Antioxid Redox Signal. 2017 Feb 10;26(5):193-206. doi: 10.1089/ars.2016.6778. Epub 2016 Sep 7. PMID 27488221
- [Background] Tang RMY, Cheah IK, Yew TSK, Halliwell B. Distribution and accumulation of dietary ergothioneine and its metabolites in mouse tissues. Sci Rep. 2018 Jan 25;8(1):1601. doi: 10.1038/s41598-018-20021-z. PMID 29371632
- [Background] Gruber J, Fong S, Chen CB, Yoong S, Pastorin G, Schaffer S, Cheah I, Halliwell B. Mitochondria-targeted antioxidants and metabolic modulators as pharmacological interventions to slow ageing. Biotechnol Adv. 2013 Sep-Oct;31(5):563-92. doi: 10.1016/j.biotechadv.2012.09.005. Epub 2012 Sep 27. PMID 23022622
- [Background] Halliwell B, Cheah I. Are age-related neurodegenerative diseases caused by a lack of the diet-derived compound ergothioneine? Free Radic Biol Med. 2024 May 1;217:60-67. doi: 10.1016/j.freeradbiomed.2024.03.009. Epub 2024 Mar 14. PMID 38492784
- [Background] Halliwell B, Tang RMY, Cheah IK. Diet-Derived Antioxidants: The Special Case of Ergothioneine. Annu Rev Food Sci Technol. 2023 Mar 27;14:323-345. doi: 10.1146/annurev-food-060822-122236. Epub 2023 Jan 9. PMID 36623925
- [Background] Wu LY, Cheah IK, Chong JR, Chai YL, Tan JY, Hilal S, Vrooman H, Chen CP, Halliwell B, Lai MKP. Low plasma ergothioneine levels are associated with neurodegeneration and cerebrovascular disease in dementia. Free Radic Biol Med. 2021 Dec;177:201-211. doi: 10.1016/j.freeradbiomed.2021.10.019. Epub 2021 Oct 19. PMID 34673145
- [Background] Cheah IK, Ng LT, Ng LF, Lam VY, Gruber J, Huang CYW, Goh FQ, Lim KHC, Halliwell B. Inhibition of amyloid-induced toxicity by ergothioneine in a transgenic Caenorhabditis elegans model. FEBS Lett. 2019 Aug;593(16):2139-2150. doi: 10.1002/1873-3468.13497. Epub 2019 Jun 30. PMID 31211853
- [Background] Wu LY, Kan CN, Cheah IK, Chong JR, Xu X, Vrooman H, Hilal S, Venketasubramanian N, Chen CP, Halliwell B, Lai MKP. Low Plasma Ergothioneine Predicts Cognitive and Functional Decline in an Elderly Cohort Attending Memory Clinics. Antioxidants (Basel). 2022 Aug 30;11(9):1717. doi: 10.3390/antiox11091717. PMID 36139790
- [Background] Cheah IK, Halliwell B. Ergothioneine, recent developments. Redox Biol. 2021 Jun;42:101868. doi: 10.1016/j.redox.2021.101868. Epub 2021 Jan 26. PMID 33558182
- [Derived] Yau YF, Cheah IK, Mahendran R, Tang RM, Chua RY, Goh RE, Feng L, Li J, Kua EH, Chen C, Halliwell B. Investigating the efficacy of ergothioneine to delay cognitive decline in mild cognitively impaired subjects: A pilot study. J Alzheimers Dis. 2024 Dec;102(3):841-854. doi: 10.1177/13872877241291253. Epub 2024 Nov 15. PMID 39544014